CLINICAL TRIAL: NCT00294164
Title: Phase 2/3, Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel-group, Dose-finding, Safety and Efficacy Trial of Subcutaneously Administered Serostim® (Mammalian Cell-derived Recombinant Human Growth Hormone, r-hGH) in the Treatment of Human Immunodeficiency Virus-associated Adipose Redistribution Syndrome (HARS)
Brief Title: Safety and Efficacy Trial of Serostim® in the Treatment of Subjects With Human Immunodeficiency Virus-associated Adipose Redistribution Syndrome (HARS)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22388
Record Dates: First submitted 2006-02-16; First posted 2006-02-20 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Human Immunodeficiency Virus-associated Adipose Redistribution Syndrome (HARS); Human Immunodeficiency Virus Infections
Keywords: Human Immunodeficiency Virus-associated Adipose Redistribution Syndrome (HARS); Human Immunodeficiency Virus Infections; recombinant human growth hormone (r-hGH); Serostim®; Placebo
MeSH Terms: interventions — Human Growth Hormone; Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Serostim® 4 mg daily (Experimental)
  Interventions: Drug: Serostim®
- Serostim® 4 mg alternate days (Experimental)
  Interventions: Drug: Serostim®; Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Serostim® — Serostim® will be administered subcutaneously (daily or given on alternate days with matched placebo), at a dose based on body weight measured at Baseline, with a maximum daily dose of 4 mg up to Week 24.
  Other Names: Recombinant human growth hormone (r-hGH)
  Arms: Serostim® 4 mg alternate days; Serostim® 4 mg daily
Drug: Placebo — Matching placebo will be administered subcutaneously (daily or given on alternate days with Serostim®), up to Week 24.
  Arms: Placebo; Serostim® 4 mg alternate days

SUMMARY:
This study is a Phase 2/3, multicenter, double-blind, randomized, parallel-group, placebo-controlled, dose-finding trial of Serostim® (mammalian cell-derived recombinant human growth hormone, r-hGH) versus placebo in subjects with human immunodeficiency virus-associated adipose tissue redistribution syndrome (HARS).

The primary study objective is to determine whether Serostim® treatment reduces adipose tissue maldistribution more effectively than placebo. The primary co-endpoints are derived from measures of visceral adipose tissue assessed by computerized tomography (CT) and the ratio of trunk; and limb fat assessed by dual-energy X-Ray absorptiometry (DXA) scans. Anthropometric measures, physical exams, quality of life assessments, serial photographs, and various laboratory measures will be used to address secondary objectives. These secondary objectives relate to the impact of Serostim® on Physician and subject assessments of change in body shape, health-related quality of life, attitude towards medication compliance, metabolic markers, fat redistribution, and safety.

On Day 1, eligible subjects will be randomized in a 1:1:1 ratio to receive daily Serostim®, Serostim® and placebo given on alternate days, or daily placebo. Serostim® doses will be based on body weight, with a maximum dose of 4 milligram (mg).

Therapy will continue for 12 weeks. Treatment will then be altered and the new treatment will be continued through Week 24. Interim Study Visits will be required at Weeks 2 and 4 (Treatment Period 1) and at Weeks 14 and 16 (Treatment Period 2). Subjects will be offered to be enrolled into a maintenance Protocol (Study 23056) at Week 24.

ELIGIBILITY:
Inclusion Criteria:

• Have an Human Immunodeficiency Virus (HIV) infection documented either by viral load as measured by polymerase chain reaction (PCR) amplification; or by the presence of HIV antibodies with confirmation by one of the following:

* Western blot
* Immunofluorescence assay
* Branched Deoxyribonucleic Acid (bDNA) signal amplification
* The presence of p24 antigen

These tests may have been performed at any time in the past, but the results must be available for review by the Serono monitor prior to randomization

* Have evidence of excess abdominal adipose deposition when measured using the following cut points:

  * Men: Waist circumference greater than 88.2 centimeter (cm) and waist/hip ratio greater than or equal to 0.95
  * Women: Waist circumference greater than 75.3 cm and waist/hip ratio greater than or equal to 0.9 (23)
* Be taking antiretroviral medication(s) which is (are) approved or is (are) available under a treatment investigational new drug (IND). The regimen must have remained stable for the 30 days prior to study entry. Subjects must also have agreed not to discontinue or to change their regimen for the duration of the study except as judged medically necessary
* Have parameter values less than the following limits:

  * Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), and amylase less than or equal to 3 times the upper limit of normal (Screening)
  * Fasting triglycerides less than or equal to 1,000 milligram per deciliter (mg/dL) (Screening)
  * Fasting glucose less than 110 mg/dL (Screening)
  * Two hour (120 minute) glucose less than 140 mg/dL (following an oral glucose load at Screening)
* Weigh greater than or equal to 36 kilogram (kg) (79.3 pound)
* Be between 18 and 60 years of age unless local law dictates different limits
* Be able and willing to comply with the protocol for the duration of the study
* Have given written informed consent
* If female, be post-menopausal or surgically sterilized (that is, have undergone tubal ligation or hysterectomy), or is

  * Using a contraceptive method such as a hormonal contraceptive, intra uterine device, diaphragm with spermicide, or condom with spermicide, for the duration of the study
  * Not pregnant or breast feeding

Exclusion Criteria:

* Have an active acquired immune deficiency syndrome (AIDS)-defining Opportunistic Infection (OI) as defined by the Center for Disease Control; or have had an untreated or suspected serious systemic infection, or persistent fever greater than or equal to 101 degree Fahrenheit (°F) (38.3 degree Celsius) during the 30 days prior to study entry
* Have any active malignancy, except for localized cutaneous Karposi's sarcoma (fewer than 10 lesions, none of which are larger than 2 cm, and not on active therapy)
* Have a central nervous system (CNS) mass or active CNS process associated with neurological findings
* Have unstable or untreated hypertension, defined as greater than or equal to 140/90 millimeter of mercury (mmHg) at the time of the Screening Visit, and/or has initiated or changed antihypertensive therapy in the 30 days prior to Day 1
* Have an acute critical illness treated in an intensive care unit, for example, due to complications following open heart or abdominal surgery, multiple accidental trauma, or acute respiratory failure
* Have any condition, which interferes with informed consent or protocol compliance including, but not limited to, active substance abuse and/or dementia
* Is unable to comply with the concomitant therapy restrictions
* Have ever been diagnosed with any of the following conditions:

  * Pancreatitis
  * Carpal tunnel syndrome (unless resolved by surgical release)
  * Diabetes mellitus
  * Angina pectoris
  * Coronary artery disease
  * Any disorder associated with moderate to severe edema (for example, cirrhosis, nephrotic syndrome, congestive heart failure, lymphedema)
* Allergy or hypersensitivity to growth hormone

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 245 (Actual)
Dates: Start 2001-03; Primary Completion 2002-05 (Actual); Study Completion 2002-05 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in absolute area of visceral adipose tissue quantified by Computerized Tomography (CT) scan at Week 12 | Baseline and Week 12
Change from Baseline in the ratio of trunk fat to limb fat quantified by Dual-Energy X-Ray Absorptiometry (DXA) scan at Week 12 | Baseline and Week 12

SECONDARY OUTCOMES:
Change from Baseline in composite sum of the visceral adipose tissue and the ratio of trunk fat to limb fat at Week 12 | Baseline and Week 12
Dorsal fat area in the transverse plane, as measured by Computerized Tomography (CT) Scan | Baseline, Week 12 and 24
Weight measured on a calibrated scale | Baseline, Week 12 and 24
Absolute values of maximal chest, waist, and hip circumference | Baseline, Week 12 and 24
Waist/hip ratio | Baseline, Week 12 and 24
Absolute value of dorsocervical fat | Baseline, Week 12 and 24
Absolute value of total body fat as quantified by DXA scan | Baseline, Week 12 and 24
Absolute value of trunk and Limb fat quantified by DXA scan | Baseline, Week 12 and 24
Absolute value of Lean body mass as quantified by DXA scan | Baseline, Week 12 and 24
Absolute concentration of serum insulin and glucose | Baseline, Week 12 and 24
Absolute concentration of fasting serum triglyceride, total cholesterol, Low density lipoprotein (LDL), High density lipoprotein (HDL) and very low density lipoprotein (VLDL) | Baseline, Week 12 and 24
High density lipoprotein (HDL)/Low density lipoprotein (LDL) ratio | Baseline, Week 12 and 24
Change from Baseline in Serial Photography Parameters of chest and abdomen at Week 12 and 24 | Baseline, Week 12 and 24
Health related Quality of life | Baseline, Week 4, 12 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Brady, M.D. MPH, Study Director — EMD Serono

REFERENCES:
- [Result] Kotler DP, Muurahainen N, Grunfeld C, Wanke C, Thompson M, Saag M, Bock D, Simons G, Gertner JM; Serostim in Adipose Redistribution Syndrome Study Group. Effects of growth hormone on abnormal visceral adipose tissue accumulation and dyslipidemia in HIV-infected patients. J Acquir Immune Defic Syndr. 2004 Mar 1;35(3):239-52. doi: 10.1097/00126334-200403010-00004. PMID 15076238
- See also: Published in J Acquir Immune Defic Syndr 35; 239-252: 2004 — http://www.jaids.com/pt/re/jaids/abstract.00126334-200403010-00004.htm
- See also: Full FDA approved prescribing information can be found here — http://www.serostim.com